CLINICAL TRIAL: NCT01811706
Title: Therapeutic Effect of Dalfampridine on Gait Incoordination in Spinocerebellar Ataxias- A Randomized, Double-blinded, Placebo-controlled, Crossover Clinical Trial
Brief Title: Dalfampridine and Gait in Spinocerebellar Ataxias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20121107; 1133511 (Other: WIRB Study Number)
Record Dates: First submitted 2013-03-06; First posted 2013-03-14 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Spinocerebellar Ataxias Type 1; Spinocerebellar Ataxias Type 2; Spinocerebellar Ataxias Type 3; Spinocerebellar Ataxias Type 6
MeSH Terms: interventions — 4-Aminopyridine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dalfampridine and then placebo (Experimental): Participant first receive Dalfampridine at an oral dose of 10mg every 12 hours, for 4 weeks. After a washout period of 2 weeks, they then receive Placebo tablet orally every 12 hours, for a 4 weeks period.
  Interventions: Drug: Dalfampridine; Drug: Placebo
- Placebo, Then Dalfampridine (Experimental): Participant first receive Placebo tablet orally every 12 hours, for a 4 weeks period. After a washout period of 2 weeks, they then receive Dalfampridine at an oral dose of 10mg every 12 hours, for 4 weeks.
  Interventions: Drug: Dalfampridine; Drug: Placebo

INTERVENTIONS:
Drug: Dalfampridine — Dalfampridine will be provided at an oral dose of 10mg every 12 hours, for 4 weeks period
  Other Names: Ampyra
Drug: Placebo — Placebo will be administered orally every 12 hours, for a 4 week period.
  Other Names: Sugar Pill

SUMMARY:
Investigators expect there will be improvement in walking speed and steadiness after taking Dalfampridine, thereby improving activities of daily living and enhancing social and occupational functions for patients with spinocerebellar ataxia.

DETAILED DESCRIPTION:
Twenty spinocerebellar ataxia patients will be randomized to receive either Dalfampridine or placebo over a total period of 10 weeks. After entering the study, patients will return every 2 weeks for evaluation. After four weeks, intervention will be stopped and patient will enter a 2-week wash out period where they do not take any drug. Then, patients will be given the opposite treatment (Dalfampridine or placebo) and this "crossover" study will be performed for another 4 weeks. Investigators expect there will be improvement in walking speed and steadiness after taking Dalfampridine, thereby improving activities of daily living and enhancing social and occupational functions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals at age 18 years or older.
* Individuals who can provide the informed consent
* Genetic confirmed definite spinocerebellar ataxias (SCA)
* Able to complete two trials of the timed 25-foot walk at screening

Exclusion Criteria:

* Patients who has severe ataxia and unable to ambulate.
* Any orthopedic condition that would affect motor performance.
* Patients with secondary ataxia from general medical disorders
* Individuals who have major psychiatric disorders that prevents compliance
* History of epilepsy
* Patients with active drug or alcohol use or dependence that would interfere with adherence to study requirements
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guangbin Xia, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: First Intervention ( 4 Weeks)
Arm/Group | Dalfampridine and Then Placebo | Placebo, Then Dalfampridine
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout ( 2 Weeks)
Arm/Group | Dalfampridine and Then Placebo | Placebo, Then Dalfampridine
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Dalfampridine and Then Placebo | Placebo, Then Dalfampridine
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 20
T25FW at screening visit [Mean (Standard Deviation); unit: second] — Timed 25-Foot Walk (T25FW): The patient is directed to one end of a marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time, in seconds, is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark.
  second | 25.5 (9.7)
SARA at screening visit [Mean (Standard Deviation); unit: point] — Scale for the assessment and rating of ataxia (SARA) is a clinical scale that is based on a semiquantitative assessment of cerebellar ataxia on an impairment level. SARA has 8 items that are related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test. SARA score ranges from 0 to 40, with higher scores indicating more severe disease.
  point | 11.1 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Timed 25 Feet Walking Test (T25FW)
Description: The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time, in seconds, is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. Baseline values are recorded twice. One was at the beginning of the intervention. The second was 2 weeks after washout period and before the second intervention.
Time Frame: Baseline and 4 weeks after Dalfampridine or placebo
Population: Patient with spinocerebellar ataxia (SCA) 1, 2, 3, or 6
Measure: Mean (Standard Deviation); unit: second
Groups:
- Dalfampridine: Participant who received Dalfampridine at an oral dose of 10mg every 12 hours for 4 weeks period.
- Placebo: Participant who received Placebo orally every 12 hours for a 4 week period.
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 19 | 19
second
  T25FW at baseline | 23.7 (10.1) | 24.4 (10.1)
  Change from baseline at 4 weeks | -1.1 (4.7) | -0.3 (4.8)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Null hypothesis is that there was no difference in change of T25FW between Dalfampridine and Placebo. The test was performed with a significant level of 0.05 (two-sided); Test type: Superiority or Other; p > 0.05, t-test, 2 sided

2. Secondary Outcome: Change in Scale of Assessment and Rating of Ataxia (SARA)
Description: Scale for the assessment and rating of ataxia (SARA) is a clinical scale that is based on a semiquantitative assessment of cerebellar ataxia on an impairment level. SARA has 8 items that are related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test. SARA score ranges from 0 to 40, with higher scores indicating more severe disease.
Time Frame: Baseline and 4 weeks after Dalfampridine or placebo
Measure: Mean (Standard Deviation); unit: point
Groups:
- Dalfampridine: Participant received Dalfampridine at an oral dose of 10mg every 12 hours, for 4 weeks period.
- Placebo: Participant received Placebo orally every 12 hours for a 4 week period.
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 19 | 19
point
  SARA at baseline | 10.0 (3.5) | 10.1 (3.3)
  Change from baseline at week 4 | 0.6 (1.5) | 0.8 (1.8)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Null hypothesis is that there was no difference in change of SARA score between Dalfampridine and Placebo. The test was performed with a significant level of 0.05 (two-sided); Test type: Superiority or Other; p > 0.05, t-test, 2 sided

3. Secondary Outcome: Biomechanical Assessment of Gait (BAG)-Stride Length
Description: Biomechanical Assessment of Gait is a sensitive, quantitative movement analysis system. Stride length was analyzed. Baseline values are recorded twice. One was at the beginning of the intervention. The second was 2 weeks after washout period and before the second intervention.
Time Frame: Baseline and 4 weeks after Dalfampridine or placebo
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 19 | 19
cm
  Sstride Length at baseline | 112.7 (29.4) | 111.8 (30.0)
  Stride Length at week 4 | 1.6 (9.4) | 4.0 (9.9)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Null hypothesis is that there was no difference in change of Stride Length on BAG between Dalfampridine and Placebo. The test was performed with a significant level of 0.05 (two-sided); Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 10 weeks per patient
Arm/Group | Dalfampridine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 7/20 | 8/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalfampridine (N=20) | Placebo (N=19)
headache (Nervous system disorders) | 3 (3) | 1 (1) — Two grade 1 headaches, and one grade 2 headache.
lethargy (Nervous system disorders) | 1 (1) | 0 (0) — grade 1
dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) — grade 3 - tooth removal
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — increased pain in the left leg
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) — grade 1
tremor (Nervous system disorders) | 0 (0) | 1 (1) — Grade 1 tremor of finger
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — grade 2
dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) — grade 2
gait disturbance (General disorders) | 1 (1) | 4 (4) — all grade 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — grade 1 - knee pain
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — grade 1
chills (General disorders) | 0 (0) | 1 (1) — grade 1
somnolence (Nervous system disorders) | 0 (0) | 1 (1) — grade 1
urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) — grade 1
blurred vision (Eye disorders) | 1 (1) | 0 (0) — grade 1 accommodation issues
voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — grade 2 - slurring of speech
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes